CLINICAL TRIAL: NCT07119970
Title: Prospective Study for the Evaluation of the Prognostic Value of NETosis Markers to Predict Thrombosis in Myeloproliferative Neoplasms With JAK2V617F Mutation (AVATARE)
Brief Title: Prognostic Value of NETosis Markers for Thrombosis During Myeloproliferative Neoplasms (AVATARE)
Acronym: AVATARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX 2023/91
Record Dates: First submitted 2025-07-01; First posted 2025-08-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Myeloproliferative Neoplasm; Myeloproliferative Disorders
Keywords: Myeloproliferative neoplasms; Thrombosis; Neutrophil extracellular traps; Neutrophils
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct oral anticoagulants (DOACs) (Experimental)
  Interventions: Biological: Additional blood sampling
- Aspirin (Active Comparator)
  Interventions: Biological: Additional blood sampling

INTERVENTIONS:
Biological: Additional blood sampling — At inclusion (T0) and at 12 months (T1), venous blood will be drawn for plasma markers of NETosis

SUMMARY:
Myeloproliferative neoplasms are hematologic diseases characterized by an increased proliferation of peripheral blood cells. The main risk of MPN is the occurrence of thrombosis. Thrombosis risk is mainly evaluated using two criteria: age and prior thrombosis. A better prediction of thrombosis risk is needed to improve prevention and treatment of MPN-associated thrombosis. The objective of the study is to evaluate the predictive value of neutrophil extracellular traps markers in thrombosis during MPN.

DETAILED DESCRIPTION:
JAK2V617F positive myeloproliferative neoplasms (MPNs) are clonal disorders of hematopoietic stem cells characterized by an increased risk of thrombosis, the main cause of morbidity and mortality in these patients. Classical risk factors for thrombosis include a prior thrombotic event and age over 60. However, these criteria are often insufficient, as some patients who receive treatment continue to experience thrombosis, while others may be overtreated based solely on age. Recent studies have highlighted the role of neutrophil extracellular traps (NETs) in thrombosis, suggesting that NETosis, the process of NET formation, contributes to the activation of hemostasis and coagulation. Increased levels of NETs have been observed in patients with MPNs, particularly those with a history of thrombosis. Aspirin has shown a potential to reduce NET formation and the occurrence of thrombosis by inhibiting platelet-triggered NETosis. This study aims to prospectively evaluate the prognostic value of NETosis markers to predict thrombosis and optimize thrombotic prevention strategies in JAK2V617F-positive MPN patients.

The AVATARE ancillary study is linked to the AVAJAK clinical trial, which compares the efficacy of aspirin versus direct oral anticoagulants (DOACs) in preventing thrombotic events. Patients included in the AVATARE study will undergo venous blood sampling at baseline (T0) and 12 months (T1) for NETosis markers, such as calprotectin and citrullinated histone H3 (H3Cit). Participants will be followed up for 24 months. Clinical data, including the occurrence of venous and arterial thrombotic events, will be collected during the study period. Blood samples will be taken at inclusion (T0) and at 12 months (T1). The progression of NETosis markers will be monitored, and their correlation with thrombotic outcomes will be assessed to understand the potential role of these markers in predicting future thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Polycythemia Vera (PV), Essential Thrombocythemia (ET), or pre-myelofibrosis (pre-MF)
* JAK2V617F mutation with an allelic burden greater than 1%
* High risk of thrombosis (age over 60 years or prior thrombotic event)
* Diagnosis of MPN within the last 12 months
* Enrollment in the AVAJAK clinical trial and the FIMBANK biobank
* Affiliation with social security
* Signed informed consent

Exclusion Criteria:

* Severe hepatic or renal insufficiency (Creatinine clearance <30ml/min)
* Patients under legal protection (guardianship or curatorship)
* Patients under heparin treatment at inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Serum calprotectin concentration | At T0 (inclusion)
  This concentration will be compared between MPN patients who develop thrombotic events during the follow-up and those who do not. The serum concentration will be measured using automated immunoturbidimetric test and the results will be analyzed to assess its association with future thrombotic events in patients with myeloproliferative neoplasms.

SECONDARY OUTCOMES:
Serum calprotectin concentration | At T1 (12 months post-inclusion)
Serum concentration of citrullinated histone H3 (H3Cit) | At T1 (12 months post-inclusion)
  This concentration will be assessed to evaluate calprotectin concentration at T1 and to compare the evolution of this marker in patients treated by direct oral anticoagulant or by aspirin.
Plasma citrullinated histone 3 concentration | At T0 (inclusion)
  This concentration will be compared between MPN patients who develop thrombotic events during the follow-up and those who do not. The plasma concentration will be measured using ELISA test and the results will be analyzed to assess its association with future thrombotic events in patients with myeloproliferative neoplasms.
Plasma citrullinated histone 3 concentration | At T1 (12 months post-inclusion)
  This concentration will be assessed to evaluate citrullinated histone 3 concentration at T1 and to compare the evolution of this marker in patients treated by direct oral anticoagulant or by aspirin.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre GUY, Principal Investigator — alexandre.guy@chu-bordeaux.fr
Locations (15):
- France (15):
  - CHU d'Angers, Service des maladies du Sang, Angers
  - CH de la Côte Basque, Service Hématologie, Bayonne
  - CHU de Bordeaux, Service Hématologie Biologique, Bordeaux
  - CHU de Bordeaux, Service Hématologie Clinique et Thérapie Cellulaire, Bordeaux
  - CHU de Brest, Service Hématologie et Hémostase Clinique, Brest
  - APHP-Hôpital Mondor, Service Hématologie Clinique et Thérapie Cellulaire, Créteil
  - CHD de Vendée, Service Onco-hématologie, La Roche-sur-Yon
  - APHP-Hôpital Bicêtre, Service Hématologie Clinique Ambulatoire, Le Kremlin-Bicêtre
  - CH de Libourne, Service Hématologie, Libourne
  - CHU de Limoges, Service Hématologie Clinique et de Thérapie Cellulaire, Limoges
  - CH des Pays de Morlaix, Service Onco-Hématologie, Morlaix
  - CHU de Nantes, Service Hématologie Clinique, Nantes
  - Hôpital Privé du Confluent, Service Hématologie, Nantes
  - APHO-Hôpital Saint-Louis, Centre d'Investigations Cliniques, Paris
  - CH de Roubaix, Service Hématologie, Roubaix

IPD SHARING:
Plan to Share IPD: No